CLINICAL TRIAL: NCT04032418
Title: Randomized Phase II Study of Pembrolizumab 200mg every12 Weeks Versus Every 3 Weeks in NSCLC With Clinical Benefit to Pembrolizumab Monotherapy: Multicenter International Study
Brief Title: Pembrolizumab Every 12 Weeks Versus Every 3 Weeks in Treating Patients With Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: i 82319; NCI-2019-04326 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); i 82319 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-07-18; First posted 2019-07-25 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (200mg pembrolizumab 3 weeks) (Active Comparator): Patients receive 200mg pembrolizumab IV over 30 minutes every 3 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab
- Arm II (200mg pembrolizumab 12 weeks) (Experimental): Patients receive 200mg pembrolizumab IV over 30 minutes every 12 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab given every 12 weeks works compared to every 3 weeks in treating patients with non-small cell lung cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving pembrolizumab every 12 weeks may provide similar disease control with fewer treatments for patients with non-small cell lung cancer when compared to every 3 weeks. Demonstrating that 12 week dosing is as effective as 3 week dosing may also have a significant impact when considering the cost required for these medications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the 1-year progression-free survival rate with 200mg pembrolizumab administered every 3 weeks compared to 200mg pembrolizumab administered every 12 weeks.

SECONDARY OBJECTIVES:

I. To assess overall survival between the two treatment groups. II. To assess the serious adverse event profiles between the two treatment groups.

EXPLORATORY OBJECTIVES:

I. To evaluate circulating biomarkers of treatment response and resistance. II. To characterize fecal microbiotic profile and to correlate those results with tumor characteristics and antitumor immune responses.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive pembrolizumab intravenously (IV) over 30 minutes every 3 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive pembrolizumab IV over 30 minutes every 12 weeks for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then every 12 weeks for at least 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2 at the time of study treatment initiation.
* Have pathologically confirmed diagnosis of non-small cell lung cancer (NSCLC). Mixed small cell lung cancer (SCLC) histology is not allowed.
* Must be eligible for treatment with pembrolizumab as standard of care (up to third line).
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L.
* Platelets >= 100 x 10^9/L.
* Hemoglobin >= 9 g/dL.
* Plasma creatinine =< 1.5 x institution upper limit of normal (ULN) or estimated glomerular filtration rate (GFR) (measured or calculated with Cockcroft and Gault formula) > 45 ml/min.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (ALT and AST =< 5 x ULN is acceptable if liver metastases are present).
* Total plasma bilirubin =< 1.5 x ULN. For patients with well documented Gilbert?s syndrome, total bilirubin =< 3 x ULN with direct bilirubin within normal range.
* Must have demonstrated complete response, partial response by Response Evaluation Criteria in Solid Tumors (RECIST) or stable disease if > 5% but less than 30% decrease from baseline total tumor burden (target lesions) to pembrolizumab at the time of randomization for study treatment.Patients with new brain metastasis isolated in the brain while on pembrolizumab monotherapy will be eligible as long as extracranial disease control fulfills the criteria otherwise (i.e. this will not be considered as disease progression for the purpose of this study).
* Must have received at least 6 months of pembrolizumab monotherapy treatment (but no more than 15 months total duration, including treatment in combination with chemotherapy prior to maintenance phase) prior to start of protocol-assigned treatment.
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Receipt of anticancer chemotherapy, other than pembrolizumab, within 6 months prior to randomization.
* Disease progression to pembrolizumab as assessed by immune related (ir)RECIST.
* Prior radiotherapy or gamma knife within 2 weeks of study treatment for non-brain metastasis. Subjects must have recovered from all radiation related toxicities.
* Active/untreated brain metastasis. Whole brain radiation or gamma knife radiosurgery performed less than 4 weeks prior to first administration of study drug. Previously treated brain metastasis allowed as long as not requiring steroids and stable on imaging at least 4 weeks after completing radiation therapy.
* Leptomeningeal involvement regardless of tumor response status.
* Tumor with mutation that is known to be sensitive to Food and Drug Administration (FDA)- approved targeted therapy.
* Patients who had pembrolizumab interrupted for more than 4 weeks for management of treatment-related adverse event.
* Currently receiving or has received high-dose systemic corticosteroids within 4 weeks prior to starting study drug for management of brain metastases, or who have not fully recovered from side effects of such treatment. Patients who are on low-dose prednisone (10 mg once daily or less) for at least 6 months for the management of other chronic disorders (e.g. chronic obstructive pulmonary disease [COPD]) is allowed. Steroids for endocrine replacement or receipt of short-course of steroids during the preceding 4 week period as supportive medication such as for drug allergy, anti-emetic, etc. is allowed.
* Had major surgery within 14 days prior to starting protocol treatment.
* Active, clinically serious infections or other serious uncontrolled medical conditions.
* Pregnant or nursing female participants.
* Any condition which in the investigator?s opinion deems the participant an unsuitable candidate to receive study drug.
* Unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
1-year progression-free survival (PFS) | Baseline to 12 months
  Measured using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Overall survival | Up to 12 months after treatment completion
  Defined as the number of months between Loading Phase enrollment and death from any cause. Analysis of overall survival between the two treatment groups will be carried forth using a log-rank test accounting for the stratification factors, including other known variables such as PD-L1 tumor proportion score, line of therapy, histology, mutation profile.
Incidence of adverse events | Up to 12 months
  Assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Will be assessed through the evaluation of grade 3 or higher toxicities deemed possibly related to treatment. Both efficacy and toxicity rates will be estimated using simple relative frequencies. The corresponding 95% confidence intervals for the estimated probabilities will be computed.

OTHER OUTCOMES:
Cox regression models in terms of treatment resistance | Up to 12 months
  Circulating biomarkers of treatment response and resistance
Length of time on treatment | Up to 12 months
  Length of time on treatment as a time varying covariate will be carried out using Cox regression models.

CONTACTS AND LOCATIONS:
Overall Officials: Grace K Dy, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States